CLINICAL TRIAL: NCT03407131
Title: Internal Fixation or Joint Replacement Therapy for Hip Fracture Patients Over 75 Years Old Combined With Multiple Internal Medicine Complications: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Internal Fixation or Joint Replacement Therapy for Aged Hip Fracture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, baoguojiang, Dean of Peking University People's Hospital, Director of department of orthopaedic surgery of Peking University, Chairman of China trauma rescue&treatment association, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUPH20171228
Record Dates: First submitted 2018-01-11; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Intertrochanteric Fractures
Keywords: Intertrochanteric fracture, Medical complications
MeSH Terms: conditions — Hip Fractures | interventions — Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint replacement (Experimental): Intertrochanteric fracture patients were treated with joint replacement surgery.The postoperative drainage volume, blood transfusion volume, intraoperative blood loss, operative time, early weight bearing time will be recorded, and postoperative pulmonary infection, urinary tract infection, bedsore incidence and postoperative functional rehabilitation will be observed.
  Interventions: Procedure: Joint replacement surgery
- Intramedullary nail fixation (Active Comparator): Intertrochanteric fracture patients were treated with intramedullary nail fixation surgery.The postoperative drainage volume, blood transfusion volume, intraoperative blood loss, operative time, early weight bearing time will be recorded, and postoperative pulmonary infection, urinary tract infection, bedsore incidence and postoperative functional rehabilitation will be observed.
  Interventions: Procedure: Intramedullary nail fixation

INTERVENTIONS:
Procedure: Joint replacement surgery — Joint replacement surgery is to replace the original joint function, so that the patient can recover the joint function as soon as possible.
  Arms: Joint replacement
Procedure: Intramedullary nail fixation — Internal fixation surgery is the stable fixation of fracture, which provides the condition for the restoration of joint function.
  Arms: Intramedullary nail fixation

SUMMARY:
To evaluate the efficacy and safety of internal fixation or arthroplasty for hip fracture patients over 75 years of age with multiple medical complications through the operation time, intraoperative bleeding, time to start weight bearing activities and other indicators.

DETAILED DESCRIPTION:
Patients will be enrolled from five study centers, each center will be free with regard to surgical indications and postoperative prescription. The unstable fractures were A2 and A3 (31 A2.2 and 3, and 31 A3.3) according to the AO classification. The investigators will use a prospective randomized approach to determine the treatment procedure for patients. The patients undergoing arthroplasty will be regarded as the experimental group and the patients who accept the intramedullary nail fixation will be regarded as the positive control group. All patients will receive consistent anticoagulant, analgesic and other therapeutic measures in the perioperative period except for the different surgical methods. The two groups will be compared in age, sex, pre-fracture place of residence, fracture type and preoperative comorbidity. The investigators will evaluate the effect and safety of the two types of operations by comparing the surgical related data, complication incidence and functional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric fractures of the femur need surgery
* Male and female, age more than 75 years old
* Combined with more than one medical complication, including hypertension, cerebral infarction, respiratory failure, renal insufficiency, coronary heart disease, diabetes, heart failure, pulmonary infection, heart rate, water and electrolyte disorders
* The patient is still able to tolerate surgery through the anaesthesia and related department assessment
* Signed written informed consent

Exclusion Criteria:

* No complications associated with internal medicine
* Mild fracture displacement and conservative treatment required
* Multiple trauma involving more than one organ system
* Known to have progressive malignant neoplasms
* It is not possible for the subjects to follow the test scheme, such as uncooperative attitudes, inability to return to the research centre for follow-up visits and inability to complete the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding related index | Three days after the operation
  Postoperative drainage volume and bleeding volume during operation（Unit: ml）

SECONDARY OUTCOMES:
Joint rehabilitation index | Three months after the operation
  Early loading time
Complication rate | Three monthes after the operation
  The incidence of postoperative lung infection, urinary tract infection, bedsore and mortality
Functional rehabilitation index | Three months after the operation
  Harris Scores of the two groups
Surgical related index | Three days after the operation
  operation time of the two groups（Unit: minutes）

CONTACTS AND LOCATIONS:
Overall Officials: Baoguo Jiang, Doctor, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided